CLINICAL TRIAL: NCT06985758
Title: Phase IV, Open-label, Single Arm, Multicenter Trial to Evaluate Pharmacokinetic Parameters of Peritoneal Diffusion and Peritoneal Diffusion Activity.
Brief Title: Pharmacokinetic Study of Rezafungin in Patients With Suspected Intra-Abdominal Candidiasis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REZAPACQ
Record Dates: First submitted 2025-04-24; First posted 2025-05-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Candidal Peritonitis
MeSH Terms: interventions — Rezafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rezafungin 400mg followed by weekly doses of intravenous Rezafungin 200mg (Experimental): Intravenous administration of a first dose of Rezafungin 400mg followed by weekly doses of intravenous Rezafungin 200mg to study the pharmacokinetic parameters of the drug.
  Interventions: Drug: Rezafungin 400mg followed by weekly doses of intravenous Rezafungin 200mg

INTERVENTIONS:
Drug: Rezafungin 400mg followed by weekly doses of intravenous Rezafungin 200mg — Intravenous administration of a first dose of Rezafungin 400mg followed by weekly doses of intravenous Rezafungin 200mg to study the pharmacokinetic parameters of the drug.
  Other Names: Rezafungin

SUMMARY:
Intra-abdominal candidiasis is the most frequent candidiasis infection after candidemia. The studies that have positioned echinocandins as the first therapeutic option in candidiasis have been carried out mainly in patients with candidemia. Peritoneal concentrations of caspofungin, micafungin and anidulafungin are clearly above the MICs of most Candida spp but are below the threshold for selection of resistant mutants, which has been argued by some researchers as a risk for the control of intra-abdominal infections with poor control of the focus and selection of resistant mutants, observed in Candida spp isolates at the peritoneal level in relation to isolates at the blood culture level.

Rezafungin, with its special pharmacokinetics, achieves higher tissue concentrations, including hepato-splenic and other abdominal organs, than the other echinocandins. Experimental studies have confirmed that the concentration of rezafungin at the level of the inflammatory focus in abdominal infections is higher than in the surrounding healthy tissue and higher than those achieved by micafungin. Finally, the biofilm activity of rezafungin is very high, clearly superior to fluconazole and possibly higher than that of other echinocandins.

DETAILED DESCRIPTION:
Intra-abdominal candidiasis is the most common candidal infection after candididaemia. Studies that have positioned echinocandins as the first therapeutic option in candidiasis have been conducted primarily in patients with candidaemia. Peritoneal concentrations of caspofungin, micafungin and anidulafungin are clearly above the MICs of most Candida spp but are below the threshold for selection of resistant mutants, which has been argued by some researchers as a risk for the control of intra-abdominal infections with poor control of the focus and selection of resistant mutants, observed in Candida spp isolates at the peritoneal level relative to isolates at the blood culture level.

Rezafungin has the characteristic of having a modified chemical structure that gives it greater stability and a prolonged half-life, allowing the drug to be administered less frequently on a weekly rather than daily basis. This results in greater clearance of candidemia and greater penetration and persistence in tissues compared to other echinocandins, and improves patient adherence to treatment.

The efficacy of Rezafungin has already been evaluated in clinical trials, and has been shown to be equal or superior to that of other echinocandins, and because it has a low incidence of cross-resistance with other antifungals, it is an appropriate choice for resistant fungal infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicion, confirmed or not, of candidiasis peritonitis or intra-abdominal infection by Candida spp. who, after having received information about the design, the purpose of the study, the possible risks that may arise from it and that they can refuse to collaborate at any time, give written consent to participate in the study.
* Be over 18 years of age
* Understand the purpose of the study and be available to perform the visits and procedures established in the protocol
* In women: negative urine pregnancy test performed in the 7 days prior to the start of study treatment in women of childbearing age and if < 2 years have passed after menopause
* Patients with signs of peritonitis or intra-abdominal infection showing refractoriness after at least 48 hours of empirical or specific antibiotherapy and in whom candidiasis infection is suspected.
* Patients with abdominal or peritoneal drainage with permeable debit that allows obtaining peritoneal samples through it.

Exclusion Criteria:

* Patients in whom there is any contraindication for use according to the established in the technical data sheet or known hypersensitivity to rezafungin or who, according to the investigator's criteria, it is not advisable to participate.
* Patients who do not present suspicion of intra-abdominal candidiasis infection or who are receiving antifungal treatment for another reason.
* Patients receiving another antifungal drug during rezafungin administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Peack Plasma Concentration (Cmax) | 7 days
  Evaluation of the ratio between Cmax, Cmin and Area Under the Rezafungin Curve in peritoneal fluid in relation to Cmax, Cmin and Area Under the Rezafungin Curve levels in blood.
Minimum Plasma Concentration (Cmin) | 7 days
  Evaluation of the ratio between Cmax, Cmin and Area Under the Rezafungin Curve in peritoneal fluid in relation to Cmax, Cmin and Area Under the Rezafungin Curve levels in blood.
Area Under the Rezafungin Curve levels in blood. | 7 days
  Evaluation of the ratio between Cmax, Cmin and Area Under the Rezafungin Curve in peritoneal fluid in relation to Cmax, Cmin and Area Under the Rezafungin Curve levels in blood.
Death curve analysis | 7 days
  Analysis of peritoneal fluid death curves in the samples per patient obtained

SECONDARY OUTCOMES:
Duration of treatment | 8 weeks
  Time in days or weeks that the treatment lasts for each patient
Overall mortality | 8 weeks
  Mortality, related or not to the treatment
Atributable mortality | 8 weeks
  Mortality related to the treatment
Blood tests | 8 weeks
  Data obtained from the performance of blood tests
Intra-abdominal cultures | 8 weeks
  Data obtained from intra-abdominal cultures
Radiology tests | 8 weeks
  Data obtained from radiology tests
Analytical tests | 8 weeks
  Data obtained from analytical tests

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Fortún Abete, MD, Principal Investigator — IRYCIS. Hospital Universitario Ramón y Cajal. Madrid, Spain.
Locations (3):
- Spain (3):
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No